CLINICAL TRIAL: NCT06055088
Title: The Effect of Hand-Foot Exercises on Peripheral Neuropathy in Women With Breast Cancer Receiving Neurotoxic Chemotherapy
Brief Title: Hand-Foot Exercises on Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-NU-678
Record Dates: First submitted 2023-09-17; First posted 2023-09-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Neuropathy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exercise with massage ball (Experimental): The exercise group will participate in home-based hand and foot exercises for 8 weeks. The exercise program will start the week the first neuropathy symptom appears and continue for 8 weeks. The exercises, which will last for 8 weeks, will be performed 3 times a day and at least 3 times a week. A detailed exercise brochure will be given to the exercise group. Patients in the massage ball group will be given a massage ball to be used in exercises.
  Interventions: Other: Hand and foot exercise
- exercise with stress ball (Experimental): The exercise group will participate in home-based hand and foot exercises for 8 weeks. The exercise program will start the week the first neuropathy symptom appears and continue for 8 weeks. The exercises, which will last for 8 weeks, will be performed 3 times a day and at least 3 times a week. A detailed exercise brochure will be given to the exercise group. Patients in the stress ball group will be given a stress ball to be used in exercises
  Interventions: Other: Hand and foot exercise
- control (No Intervention): No intervention will be applied to the patients in the control group during the follow-up period, only data collection forms will be applied.

INTERVENTIONS:
Other: Hand and foot exercise — The exercise group will participate in home-based hand and foot exercises for 8 weeks. The exercise program will start the week the first neuropathy symptom appears and continue for 8 weeks. The exercises, which will last for 8 weeks, will be performed 3 times a day and at least 3 times a week.
  Patients in the massage ball group will be given a massage ball to be used in exercises. Patients in the stress ball group will be given a stress ball to be used in exercises.
  Arms: exercise with massage ball; exercise with stress ball

SUMMARY:
This study will be conducted to compare the effects of hand and foot exercises on peripheral neuropathy and quality of life in breast cancer patients taking taxanes

DETAILED DESCRIPTION:
İntroduction: New evaluation and care strategies for symptom control are gaining importance due to the increasing prevalence of cancer, expansion of chemotherapy indications, and the development of new chemotherapeutic agents with side effects such as peripheral neuropathy and pain. In the literature review, although there are studies evaluating the effects of neuropathic pain, neuropathy on quality of life and daily living activities, it was determined that there are a very limited number of studies on reducing chemotherapy-induced neuropathy. Simple, at-home exercises to prevent neuropathy can be done daily in a short period of time and do not require special equipment. These exercises may serve as an alternative therapy to improve quality of life by reducing pain in people with neuropathy.

Purpose: This study will be conducted to compare the effects of hand and foot exercises on peripheral neuropathy and quality of life in breast cancer patients taking taxanes.

Method: This study will be conducted using a randomized controlled research design. The research sample will consist of 84 women with breast cancer receiving chemotherapy in the chemotherapy unit of a training and research hospital. Research data will be collected using the Introductory Information Form, Visual Analog Questionnaire (VAS), National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0) -Peripheral Neuropathy, EORTC QLQ-CIPN 20. The exercise program will start the week the first neuropathy symptom appears and continue for 8 weeks. Data will be collected in two time periods: the week of starting exercise (T1) and the 8th week after exercise (T2).

Conclusion: It is thought that home-based, simple exercise practices will reduce neuropathy symptoms and improve the quality of life in women with breast cancer receiving neurotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* The age of 18-80 years
* Clinical diagnosis of breast cancer
* Must be able to read and speak Turkish
* Must be the first time the taxane group receives chemotherapy
* Must be have at least grade 1 neuropathy according to CTCAE
* Must agree to participate in the study

Exclusion Criteria:

* Presence of peripheral neuropathy conditions not caused by chemotherapy [tumor compression, nutritional disorders, infections, neurological diseases such as stroke, diabetes, etc.]
* Skin infection, scar tissue, inflammation, or cuts on the hands or feet
* Neuropsychiatric disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0(NCI-CTCAE v5.0): | 8 week
  NCI-CTCAE v.5.0 publishes standardized definitions for known adverse events and defines the severity of organ toxicities for patients receiving cancer treatment. In NCI-CTCAE, the severity of chemotherapy-related peripheral neuropathy is divided into two: motor and sensory peripheral neuropathy, and the severity of complaints that interfere with patients' daily life and personal care is questioned.
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy (EORTC QLQ- CIPN 20) | 8 week
  It reveals the effects of chemotherapy-related peripheral neuropathy symptoms and the functional limitations caused by these symptoms on patients. The scale includes sensory (tingling, numbness, pain, unsteadiness when walking or standing, distinguishing temperature and hearing), motor (cramps, writing, grasping small objects, weakness) and autonomic (dizziness after changing position, vision, erectile dysfunction). It has 3 subscales: The 20 items in the scale are Likert type and the answers are evaluated by giving 1 point at all, 2 a little bit, 3 points a lot, 4 points a lot. High scores from these sections indicate more symptoms and problems, and low scores indicate fewer symptoms and problems.
Visual Analog Scale (VAS) | 8 week
  Visual Analog Scale (VAS) pain score was evaluated as "no pain" (score = 0) and "worst pain" (score = 10).

CONTACTS AND LOCATIONS:
Overall Officials: Neşe Uysal, Study Director — Amasya U
Locations (1):
- Health Science University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Uysal N, Unal Toprak F. The effect of hand and foot exercises on peripheral neuropathy and quality of life in women with breast cancer: a randomized controlled trial. Support Care Cancer. 2025 Jan 8;33(2):83. doi: 10.1007/s00520-025-09145-x. PMID 39779496